CLINICAL TRIAL: NCT05163860
Title: Implications of Family Relationships on Nutrition and Health Behaviors in Transgender and Gender Diverse (TGGD) Youth and Young Adults
Brief Title: Family Relationships and Nutrition in TGGD Youth and Young Adults
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Sarah Bostic, B.S., Graduate Student, St. Louis University
Other Study IDs: 31659
Record Dates: First submitted 2021-11-13; First posted 2021-12-20 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Family Relations; Nutrition Disorders; Health Behavior; Transgenderism
Keywords: Youth; Young Adult; Transgender; Gender Diverse; Nutrition; Health Behavior; Family Relationship; Trans; Eating Disorder; Food Insecurity; Malnutrition; Physical Activity
MeSH Terms: conditions — Nutrition Disorders; Health Behavior; Transsexualism; Feeding and Eating Disorders; Malnutrition; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Youth: TGGD youth age 12-17 will answer a survey regarding demographics (gender identity, sex assigned at birth, age, religion, degree of religiosity, degree of family religiosity, degree of conservatism/liberalism, degree of family conservatism/liberalism, ethnicity), age at which they revealed their gender identity, family gender environment (FGE), eating disorder risk (ADO-BED, previous Eating Disorder diagnosis), food insecurity (HVS), perceived support of healthy eating and physical activity (SheL), risk taking behavior (ARQ), adequacy of physical activity (PACE+), bodyweight (BMI, BMI%ile, %mBMI), and previously diagnosed psychiatric and neurodevelopmental disorders
  Interventions: Other: Survey
- Young Adults: TGGD young adults age 18-25 will answer a survey regarding demographics (gender identity, sex assigned at birth, country of residence, ethnicity, age, religion, degree of religiosity, degree of family religiosity, degree of conservatism/liberalism), age at which they revealed their gender identity, family gender environment (FGE), eating disorder risk (SCOFF, ADO-BED, previous ED diagnosis), food insecurity (HVS), perceived support of healthy eating and physical activity (SheL), risk taking behavior (RRBQ), bodyweight (BMI), malnutrition risk (MST), and previously diagnosed psychiatric and neurodevelopmental disorders.
  Interventions: Other: Survey
- Parents: Parents of TGGD youth will answer a survey with information regarding demographics (religion, degree of religiosity, degree of conservatism/liberalism, country of residence, ethnicity, gender identity, sex assigned at birth, sexual orientation, education, marital status, household size, income), anxiety (GAD-7), depression (PHQ-9), family gender environment (FGE), food insecurity (HVS), height and bodyweight (BMI).
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Participants will complete an online survey.

SUMMARY:
The purpose of this study is to assess how family relationships are related to health and nutrition behaviors among transgender and gender diverse youth and young adults.

DETAILED DESCRIPTION:
The study is recruiting the following populations: parents of transgender and gender diverse youth, transgender and gender diverse young adults, and transgender and gender diverse youth. Participants over the age of 18 will be recruited via Amazon Mechanical Turk (MTurk), and youth participants will be recruited via parent referral. Age and role-appropriate surveys will be administered to the three distinct populations. A waiver of written consent for participation will be used per survey protocol. After participants receive a recruitment statement about the study and the potential risks, willing participants will take a 10-20 minute survey to provide data regarding demographics, height and weight, food habits, physical activity, food security, health support, risk-taking behaviors, past health diagnoses, and family environment. No personal identifiers will be collected and all responses will remain confidential. Our main question is whether family acceptance of a transgender or gender diverse (TGGD) youth and young adults is related to health, nutrition, and risk-taking behaviors.

ELIGIBILITY:
Inclusion Criteria:

TGGD Young Adults:

* 18 to 25 years of age
* Self-identify as transgender or gender diverse
* A resident of the United States of America or Canada
* English speaking.

Parent of TGGD Youth

* A parent of a 12-17 year old TGGD youth
* A resident of the United States of America or Canada
* English speaking
* Have a child that self-identifies as transgender or gender diverse

TGGD Youth

* 12 to 17 years of age
* Self-identify as transgender or gender diverse
* A resident of the United States of America or Canada
* English speaking

Exclusion Criteria:

TGGD Young Adults

* Less than 18 years of age or greater than 25 years of age
* Self-identify as cis-gender
* Not a resident of the United States of America or Canada
* Non-english speaking

Parent of TGGD Youth:

* Parents of children that are less than 12 years of age or greater than 17 years of age
* Not a resident of the United States of America or Canada
* Non-english speaking
* Does not identify as a parent of a TGGD child

TGGD Youth

* Less than 12 years of age or greater than 17 years of age
* Does not self-identify as transgender or gender diverse
* Not a resident of the United States of America or Canada
* Non-english speaking

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants either identify as transgender or gender diverse themselves or are the parent of a child who identifies as transgender or gender diverse.
Study Population: TGGD Young Adults: Participants are ages 18 to 25 years, resident of the US or Canada, speak English, can be of any ethnicity or socio economic status and will self-identify as transgender or gender diverse.
  Parents of TGGD Youth: Participants are ages 18 to 90 years, resident of the US or Canada, speak English, can be of any ethnicity, socio economic status, or gender, and have a child who self-identifies as transgender or gender diverse.
  TGGD Youth: Participants are ages 12-17 years, resident of the US or Canada, speak English, can be of any ethnicity or socio economic status and will self-identify as transgender or gender diverse.
Sampling Method: Non-Probability Sample
Enrollment: 714 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Family Gender Environment measures of TGGD Youth, TGGD Young Adults, and Parents of TGGD Youth | 10-20 minute survey completed at one point within the 1 month recruitment period.
  For TGGD Youth, Young Adults, and Parents, the Family Gender Environment (FGE) questionnaire will measure family acceptance. The questionnaire has 3 parts. Part 1 has a minimum score of 0 and maximum of 57; high scores on part 1 indicate family acceptance. Part 2 has a minimum score of 0 and maximum of 60. A lower score for part 2 indicates greater family acceptance. Part 3 is scored with answers to questions 1, 3, and 6 with a combined minimum of 0 and maximum of 9; a lower score indicating higher family acceptance. Questions 2, 4, and 5 have a minimum of 0 and maximum of 9; a higher score indicating higher family acceptance.
Prevalence of Food Insecurity in TGGD Youth, TGGD Young Adults, and Parents of TGGD Youth | 10-20 minute survey completed at one point within the 1 month recruitment period.
  The Hunger Vital Sign (HVS) is a validated, 2 question screening tool. A response of "often true" or "sometimes true" to either or both questions indicates a positive screen for food insecurity.
Prevalence of Support of Healthy Eating and Physical Activity in TGGD Youth and TGGD Young Adults | 10-20 minute survey completed at one point within the 1 month recruitment period.
  The Support for Healthy Lifestyle (SheL) Family Questionnaire is a 20 question measure with 3 outcomes: Healthy Eating Support, Physical Activity Support, and Hypocritical Control. Each section has a minimum score of 0 and maximum score of 4. A higher calculated score indicates greater support for a healthy lifestyle. A higher total score indicates greater support.
Prevalence of Risk Taking Behavior in TGGD Youth and TGGD Young Adults | 10-20 minute survey completed at one point within the 1 month recruitment period.
  For TGGD Youth, risk taking behavior is measured with the Adolescent Risk Taking Questionnaire (ARQ), a 28-item measure. Participants rate their behaviors on a 5-point scale, 0-4. Minimum score of 0 and maximum score of 112. Responses are summed and greater scores reflect greater perceptions of risk and greater engagement in risky behavior.
  For TGGD Young Adults, risk taking behavior is measured with the Risk and Reckless Behavior Questionnaire (RRBQ), an 18-item measure. Participants indicate frequency of engagement in behaviors in the last year, ranging from zero times to 100+ times. Scores are summed for a total score with higher numbers indicating greater risk taking behaviors.
Physical Activity Adequacy in TGGD Youth | 10-20 minute survey completed at one point within the 1 month recruitment period.
  The Patient-Centered Assessment and Counseling for Exercise plus Nutrition (PACE+) is a 2-item measure. Participants indicate the number of active days in a week with minimum 0 and maximum 7. The measure is scored by summing the responses. A score less than 5 indicates the participant is not meeting physical activity guidelines.
Body Mass Index of TGGD Youth and TGGD Young adults | 10-20 minute survey completed at one point within the 1 month recruitment period.
  Participants will respond with their height and weight, and their Body Mass Index (BMI) will be calculated (kg/m^2). Classification will be determined by Center for Disease Control guidelines for BMI. Underweight (less than 18.5), Normal (18.5-25), Overweight (25-<30), Obese (30+).
Body Mass Index Percentile of TGGD Youth | 10-20 minute survey completed at one point within the 1 month recruitment period.
  Body Mass Index Percentile (BMI%ile) evaluates growth in youth age 2-20 years. It expresses BMI for age as a percentile obtained from the Center for Disease Control graph. https://www.cdc.gov/healthyweight/assessing/bmi/childrens_bmi/about_childrens_bmi.html#percentile Participants will respond with their height and weight, and their Body Mass Index (BMI) will be calculated (kg/m^2). Classification will be determined by CDC guidelines; <5th %ile underweight, 5-85th %ile healthy, 85-95th %ile overweight, equal to or over 95th %ile obese.
Percent Median Body Mass Index for TGGD Youth | 10-20 minute survey completed at one point within the 1 month recruitment period.
  Percent Median Body Mass Index (%mBMI) is used as a comparative standard for BMI of youth age 10-19. https://www.who.int/data/gho/data/indicators/indicator-details/GHO/prevalence-of-overweight-among-children-and-adolescents-bmi-1-standard-deviations-above-the-median-(crude-estimate)-(-)
  %mBMI is calculated by comparing the BMI of the child to the median BMI for children their age, regardless of gender.
Malnutrition Risk in TGGD Young Adults | 10-20 minute survey completed at one point within the 1 month recruitment period.
  The Malnutrition Screening Tool (MST) is a 3-item measure that screens for malnutrition. Minimum value is 0 and maximum is 7. A score of 0-1 indicates no risk for malnutrition, and a score of 2 or more indicates risk for malnutrition.
Eating Disorder Risk in TGGD Youth and Young Adults | 10-20 minute survey completed at one point within the 1 month recruitment period.
  For TDDG Youth, a "yes" response to previously diagnosed eating disorder question indicates an eating disorder. The Adolescent Binge Eating Disorder Questionnaire (ADO-BED); min value 0 and max 10. High scores indicate increased risk. Positive answers to questions 1 or 2 with 6 or more positive answers to additional questions are high risk. Participants with 3 or less positive answers are low risk.
  For TGGD Young Adults, a "yes" response to previously diagnosed eating disorder question indicates an eating disorder. The Adolescent Binge Eating Disorder Questionnaire (ADO-BED) minimum value is 0 and maximum value is 10. Higher scores indicate increased risk. Positive answers to questions 1 or 2 and 6 or more positive answers to the 8 additional questions are high risk. 3 or less positive answers are low risk. The Sick, Control, One, Fat, Food, (SCOFF) Questionnaire; minimum value of 0 and maximum value of 5. A score 2 indicates a likely anorexia nervosa or bulimia nervosa.
Prevalence of Anxiety in Parents of TGGD Youth | 10-20 minute survey completed at one point within the 1 month recruitment period.
  The Generalized Anxiety Disorder-7 Questionnaire (GAD-7) total score for the 7 items ranges from 0-21. 0-4 indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety.
Prevalence of Depression in Parents of TGGD Youth | 10-20 minute survey completed at one point within the 1 month recruitment period.
  The Patient Health Questionnaire (PHQ-9) screens for severity of depression. The 9 item measure has selections from 0 "not at all" to 3 "nearly every day" and a total minimum score of 0 and maximum score of 27. Higher PHQ scores are associated with decreased functional states and increased symptom-related difficulties.
Prevalence of Psychiatric and Neurodevelopmental Disorders in TGGD Young Adults | 10-20 minute survey completed at one point within the 1 month recruitment period.
  Describe prevalence of neurological disorders in the population by having the participants select previous diagnoses from a list of conditions.
Compare Parent and Youth Reports of Family Environment, Food Insecurity, and Weight | 10-20 minute survey completed at one point within the 1 month recruitment period.
  Compare reports of family environment (FGE), food insecurity (HVS), and weight (BMI%ile, BMI, %mBMI) between parents of TGGD youth and TGGD youth.
Parent of TGGD Youth Demographics | 10-20 minute survey completed at one point within the 1 month recruitment period.
  Describe the parent of TGGD youth sample with data on demographics (religion, degree of religiosity, degree of conservatism/liberalism, country of residence, ethnicity, gender identity, sex assigned at birth, sexual orientation, education, marital status, household size, income).
TGGD Youth and TGGD Young Adult Demographics | 10-20 minute survey completed at one point within the 1 month recruitment period.
  Describe the TGGD youth and TGGD young adult sample with data on demographics (gender identity, sex assigned at birth, country of residence, ethnicity, age, religion, degree of religiosity, degree of family religiosity, degree of conservatism/liberalism).

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Linsenmeyer, Ph.D., Study Chair — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
We will not make Individual Participant Data available to other researchers.